CLINICAL TRIAL: NCT06982521
Title: A Phase 3 Open-Label Randomized Study Assessing the Efficacy and Safety of RLY-2608 + Fulvestrant Versus Capivasertib + Fulvestrant as Treatment for PIK3CA-mutant Hormone Receptor Positive, Human Epidermal Growth Factor Receptor 2 Negative (HR+/HER2-) Locally Advanced or Metastatic Breast Cancer Following Recurrence or Progression On or After Treatment With a CDK4/6 Inhibitor
Brief Title: Phase 3 Study of RLY-2608 + Fulvestrant vs Capivasertib + Fulvestrant as Treatment for Locally Advanced or Metastatic PIK3CA-mutant HR+/HER2- Breast Cancer
Acronym: ReDiscover-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Relay Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RLY-2608-102
Record Dates: First submitted 2025-05-08; First posted 2025-05-21 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-09

CONDITIONS: PIK3CA Mutation; HER2- Negative Breast Cancer; Hormone Receptor Positive Tumor; Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — capivasertib; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RLY-2608 + fulvestrant (Experimental): RLY-2608 + fulvestrant combination for participants with HR+/HER2- advanced breast cancer
  Interventions: Drug: RLY-2608; Drug: Fulvestrant
- capivasertib + fulvestrant (Active Comparator): capivasertib + fulvestrant combination for participants with HR+/HER2- advanced breast cancer
  Interventions: Drug: Capivasertib; Drug: Fulvestrant

INTERVENTIONS:
Drug: RLY-2608 — 400 mg orally BID administered daily on a 28-day treatment cycle
  Arms: RLY-2608 + fulvestrant
Drug: Capivasertib — 400mg orally BID administered on an intermittent weekly dosing schedule. Patients will dose on Days 1 through 4 each week of a 28-day treatment cycle
  Other Names: TRUQAP
  Arms: capivasertib + fulvestrant
Drug: Fulvestrant — 500 mg intramuscularly administered on Cycle 1 Day 1, Day 15, and Day 1 of each subsequent cycle (28-day treatment cycle)
  Other Names: Faslodex

SUMMARY:
This is a global, multicenter, open-label, randomized Phase 3 study comparing the efficacy and safety of RLY-2608 + fulvestrant to capivasertib + fulvestrant for the treatment of patients with HR+/HER2- ABC with PIK3CA mutation following recurrence or progression on or after treatment with a CDK4/6 inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Patient has ECOG performance status of 0-1
* One or more known primary oncogenic PIK3CA mutation(s)
* Adult females, pre- and/or post-menopausal, and adult males. Pre-menopausal (and peri-menopausal) women can be enrolled if amenable to treatment with a gonadotropin-releasing hormone (GnRH) agonist. Patients are to have commenced treatment with a GnRH agonist at least 4 weeks prior to randomization and must be willing to continue on it for the duration of the study.
* Histologically or cytologically confirmed diagnosis of HR+/HER2- locally advanced or metastatic breast cancer (ABC) with radiological or objective evidence of recurrence or progression; locally advanced disease must not be amenable to resection with curative intent
* Measurable disease per RECIST v1.1 or evaluable bone-only disease.
* Must have radiological evidence of progression on or after previous treatment for HR+/HER2- ABC with:

  1. At least 1 and no more than 2 lines of endocrine therapy (ET) in the (neo)adjuvant setting with recurrence on or within 12 months of completion or in the ABC setting
  2. 1 prior line of CDK4/6 inhibitor therapy in one of the following settings:

     1. CDK4/6 inhibitor + ET in the ABC setting
     2. CDK4/6 inhibitor therapy in the adjuvant setting if progression occurred during or within 12 months of completion of adjuvant CDK4/6 inhibitor with ET
     3. Patients who progressed during or within 12 months of completion of adjuvant CDK4/6 inhibitor and after receiving CDK4/6 inhibitor therapy in the advanced setting are considered to have had >1 prior line of CDK4/6 inhibitor and are not eligible

Exclusion Criteria:

* Prior treatment with any of the following:

  1. CDK2 or selective CDK4 inhibitors or any investigational therapies targeting cyclin dependent kinases
  2. PIK3, AKT, or mTOR inhibitors or any agent whose mechanism of action is the inhibit the PIK3/AKT/mTOR pathway
  3. Immunotherapy
  4. Antibody drug conjugates
* Type 1 diabetes, or Type 2 diabetes requiring antihyperglycemic medication, or fasting plasma glucose ≥ 140 mg/dL, or glycosylated hemoglobin (HbA1c) ≥7.0% (≥ 53 mmol/mol).
* Clinically significant, uncontrolled cardiovascular disease
* Any factors that increase the risk of QTc prolongation or risk of arrhythmic events
* Known active uncontrolled or symptomatic CNS metastases associated with progressive neurological symptoms or requiring ongoing corticosteroids or anticonvulsants for symptomatic control
* Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease
* History of hypersensitivity to fulvestrant or drugs in a similar class as fulvestrant, RLY-2608, or capivasertib, including their excipients
* Known activating AKT mutations, loss-of-function PTEN mutations, or loss of PTEN expression resulting in oncogenic pathway activation downstream of PI3K

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) within the overall and kinase population by blinded independent central review (BICR) | The time from date of randomization until radiographic progression per RECIST v1.1, or death due to any cause, up to approximately 77 months

SECONDARY OUTCOMES:
Overall Survival (OS) within the overall and kinase populations | The time from randomization to the date of death by any cause, up to approximately 77 months
PFS by Investigator within the overall and kinase populations | The time from date of randomization until radiographic progression per RECIST v1.1, or death due to any cause, up to approximately 77 months
Objective Response Rate (ORR) within the overall and kinase populations | Up to approximately 77 months
Duration of Response (DOR) within the overall and kinase populations | Up to approximately 77 months
Clinical Benefit Rate (CBR) within the overall and kinase populations | Up to approximately 77 months
Occurrence/frequency of Adverse Events (AEs) and its relationship to the study drugs (safety and tolerability) within the overall and kinase populations | Up to approximately 77 months
Plasma concentrations of RLY-2608 (and its metabolites as appropriate) | Approximately every 2 weeks in Cycle 1 (4-week cycle) and during Cycles 2 and 3
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (EORTC QLQ-C30) scale/item scores including change from baseline and time to deterioration within overall and kinase populations | Up to approximately 77 months
EORTC Quality of Life Questionnaire Breast Cancer-Specific Module (EORTC QLQ-BR23) scale/item scores including change from baseline and time to deterioration within the overall and kinase populations | Up to approximately 77 months
Health state utility data for economic evaluation by EQ-5D-5L health state utility index within the overall and kinase populations | Up to approximately 77 months

CONTACTS AND LOCATIONS:
Locations (56):
- United States (42):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - City of Hope, Duarte, California
  - Stanford University School of Medicine, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Medical Oncology Hematology Consultants, Newark, Delaware
  - Florida Cancer Specialists, Fort Myers, Florida
  - Cancer Care Centers of Brevard, Palm Bay, Florida
  - Rush Medical College, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Community Health Network, Indianapolis, Indiana
  - University of Kansas Medical Center, Westwood, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Johns Hopkins Medicine - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Profound Research LLC, Royal Oak, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - NYU Langone Cancer Center, New York, New York
  - Mount Sinai, New York, New York
  - Columbia University Herbert Irving Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology Central/South, Austin, Texas
  - Texas Oncology DFW, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - Baylor Scott and White Research Institute, Temple, Texas
  - Huntsman Cancer Center, University of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - University of Wisconsin, Madison, Wisconsin
- Ballarat Oncology & Haematology Service, Wendouree, Victoria, Australia
- Belgium (2):
  - CHU-UCL Namur, Site Sainte-Elisabeth, Namur
  - Vitaz, Campus Sint-Niklaas, Sint-Niklaas
- CEON+ Pesquisas, São Caetano do Sul, São Paulo, Brazil
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Sygehus Sønderjylland, Sønderborg
- Centre Leon Berard, Lyon, France
- Azienda Ospedaliera Universitaria Careggi, Florence, Italy
- Radboud UMC, Nijmegen, Netherlands
- Spain (4):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Beata Maria Ana/IOB Madrid, Madrid
  - Clinica Universidad de Navarra, Madrid
- Taipei Veterans General Hospital, Taipei, Taiwan